CLINICAL TRIAL: NCT03913130
Title: An Open-Label, Extension Study to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetics of QR-110 in Subjects With Leber's Congenital Amaurosis (LCA) Due to the c.2991+1655A>G Mutation (p.Cys998X) in the CEP290 Gene
Brief Title: Extension Study to Study PQ-110-001 (NCT03140969)
Acronym: INSIGHT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated [Study prematurely terminated due to sponsor decision for reasons unrelated to safety]
Sponsor: Laboratoires Thea (Industry)
Collaborators: Sepul Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PQ-110-002; 2018-003500-40 (EudraCT Number)
Record Dates: First submitted 2019-02-21; First posted 2019-04-12 (Actual); Results first posted 2023-01-04 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Leber Congenital Amaurosis 10; Blindness; Leber Congenital Amaurosis; Vision Disorders; Sensation Disorders; Neurologic Manifestations; Eye Diseases; Eye Diseases, Hereditary; Eye Disorders Congenital; Retinal Disease
Keywords: LCA10; CEP290; p.Cys998X; c.2991+1655A>G; Leber's Congenital Amaurosis; Antisense oligonucleotide; RNA therapy
MeSH Terms: conditions — Leber Congenital Amaurosis 10; Blindness; Leber Congenital Amaurosis; Vision Disorders; Sensation Disorders; Neurologic Manifestations; Eye Diseases; Eye Diseases, Hereditary; Eye Abnormalities; Retinal Diseases; Meckel Syndrome, Type 4; Optic Atrophy, Hereditary, Leber

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug QR-110 (Experimental): First treated eye: maintenance dose every 6 months, intravitreal administration Contralateral eye: loading dose followed by maintenance dose, every 6 months, intravitreal administration
  Interventions: Drug: QR-110

INTERVENTIONS:
Drug: QR-110 — First treated eye: maintenance dose every 6 months, intravitreal administration Contralateral eye: loading dose followed by maintenance dose, every 6 months, intravitreal administration

SUMMARY:
Subjects completing participation in study PQ-110-001 (EudraCT 2017-000813-22 / NCT03140969) will be given the opportunity to enroll into the extension study for continued dosing if available data support current and/or future benefits for the subject. Study PQ-110-002 will provide long-term safety, tolerability, pharmacokinetic (PK), and efficacy data of QR-110.

DETAILED DESCRIPTION:
Subjects completing participation in study PQ-110-001 (EudraCT 2017-000813-22 / NCT03140969) will be given the opportunity to enroll into the extension study for continued dosing if available data support current and/or future benefits for the subject.

Subjects will be given the opportunity to enroll into this extension study for continued dosing if available data support current and/or future benefits for the subject. The Investigator, in consultation and agreement with the Medical Monitor, will decide on enrollment of each individual subject, as well as on dosing of the first treated eye and treatment initiation of the contralateral eye. Continued subject treatment in this study is desirable, but cannot be guaranteed, since it will depend on the risks and benefit of further treatment on a case-by-case basis, as discussed and agreed upon with the Medical Monitor.

The contralateral eye and the first treated eye will be injected 3 months apart. The injection interval of 3 months between both eyes will limit burden for the subjects, with a 3 month-visit frequency during the course of the study. This between-eye interval could be adapted if safety data are supportive, and for logistic reasons, and in agreement with the Medical Monitor.

The same safety monitoring protocol and efficacy assessments will apply to both eyes.

QR-110 will be administered via intravitreal (IVT) injection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed participation in the study PQ-110-001 and who may derive benefit from continued treatment with QR 110, as assessed by the Investigator, in consultation with the Medical Monitor
* Persistence of detectable outer nuclear layer (ONL) in the area of the macula in the opinion of the Investigator, as determined by OCT.
* Clear ocular media and adequate pupillary dilation to permit good quality retinal imaging, as assessed by the Investigator.
* An adult (≥ 18 years) willing and able to provide informed consent for participation OR a minor (6 to < 18 years) with a parent or legal guardian willing and able to provide written permission for the subject's participation prior to performing any study related procedures, and pediatric subjects able to provide age-appropriate assent for study participation.
* Female subjects who have reached menarche and male subjects must either practice true abstinence in accordance with their preferred and usual lifestyle, or agree to use acceptable, highly effective methods of contraception for up to 3 months following their last dose QR-110. Acceptable methods of contraception are defined in the protocol. Women of non-childbearing potential may be included without the use of adequate birth control, provided they meet the criteria in the protocol.

Exclusion Criteria:

* Any contraindication to IVT injection according to the Investigator's clinical judgment and international guidelines (Avery 2014).
* Safety issue during study PQ-110-001 that may compromise subject safety when continued dosing, as determined by the Investigator, and in consultation with the Medical Monitor.
* Any ocular or systemic disease or condition (including medications and laboratory test abnormalities) that could compromise subject safety or interfere with assessment of efficacy and safety, as determined by the Investigator and in consultation with the Medical Monitor.
* Pregnant or breast-feeding female.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sepul Bio Chief Medical Officer, Study Director — Sepul Bio
Locations (3):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Scheie Eye Institute, University of Pennsylvania, Philadelphia, Pennsylvania
- Ghent University Hospital and Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug QR-110
Started | 9
Completed | 8
Not Completed | 1
Not completed — Sponsor Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Drug QR-110
Number analyzed (Participants) | 9
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age (Mean) | 24.7 (12.7)
Age, Customized [Median (Full Range); unit: Years]
  Age (Median) | 23.0 [10 to 45]
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 3
  >= 18 Years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Weight (Mean) [Mean (Standard Deviation); unit: kg] | 64.26 (23.19)
Weight (Median) [Median (Full Range); unit: kg] | 61.55 [40.1 to 111.2]
Height (Mean) [Mean (Standard Deviation); unit: cm] | 164.9 (11.8)
Height (Median) [Median (Full Range); unit: cm] | 166.3 [145 to 183]
BMI (Mean) [Mean (Standard Deviation); unit: kg/m2] | 23.02 (5.20)
BMI (Median) [Median (Full Range); unit: kg/m2] | 21.89 [17.2 to 33.1]
Genotype [Count of Participants; unit: Participants]
  Compound Heterozygous | 8
  Homozygous | 1

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Ocular AEs
Description: Frequency of ocular adverse events (AEs)
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Drug QR-110
Number analyzed (Participants) | 9
Participants | 7

2. Primary Outcome: Frequency of Non-ocular AEs
Description: Frequency of non-ocular AEs
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Drug QR-110
Number analyzed (Participants) | 9
Participants | 6

3. Secondary Outcome: Change in BCVA in First Treated Eye
Description: Change in Best Corrected Visual Acuity (BCVA) in First Treated Eye
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Drug QR-110
Number analyzed (Participants) | 7
logMAR | 0.03 (0.17)

4. Secondary Outcome: Change in Mobility Course Score
Description: Change in Mobility course score
Time Frame: 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Change in Photoreceptor Outer Segment Layer Thickness
Description: Change in photoreceptor outer segment layer thickness by Optical Coherence Tomography (OCT)
Time Frame: 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Change in OCI
Description: Change in Oculomotor Instability (OCI)
Time Frame: 24 months
Reporting Status: Not Posted

7. Secondary Outcome: Change in FST Blue
Description: Change in Full-Field Stimulus Testing (FST) - blue stimuli
Time Frame: 24 months
Reporting Status: Not Posted

8. Secondary Outcome: Change in FST Red
Description: Change in Full-Field Stimulus Testing (FST) - red stimuli
Time Frame: 24 months
Reporting Status: Not Posted

9. Secondary Outcome: Change in VFQ-25
Description: Change in Visual Function Questionnaire-25 (VFQ-25) score (adult subjects)
Time Frame: 24 months
Reporting Status: Not Posted

10. Secondary Outcome: Change in CVAQ
Description: Change in Cardiff Visual Ability Questionnaire for Children (CVAQC) score (pediatric subjects)
Time Frame: 24 months
Reporting Status: Not Posted

11. Secondary Outcome: Change in PLR
Description: Change in Pupillary Light Reflex (PLR) (latency and amplitude)
Time Frame: 24 months
Reporting Status: Not Posted

12. Secondary Outcome: Change in NIRAF
Description: Change in Near Infrared AutoFluorescence (NIRAF)
Time Frame: 24 months
Reporting Status: Not Posted

13. Secondary Outcome: Change in BCVA in Treated Contralateral Eye
Description: Change in Best Corrected Visual Acuity (BCVA) in Treated Contralateral Eye
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Drug QR-110
Number analyzed (Participants) | 5
logMAR | -0.11 (0.23)

14. Secondary Outcome: Change in BCVA in Non-Treated Contralateral Eye
Description: Change in Best Corrected Visual Acuity (BCVA) in Non-Treated Contralateral Eye
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Drug QR-110
Number analyzed (Participants) | 2
logMAR | 0.05 (0.21)

ADVERSE EVENTS:
Time Frame: Any event/condition noted once the subject receives their first dose of study drug in the contralateral eye will be captured as an AE. All AEs and SAEs regardless of attribution will be collected until at least 3 months following the last administration of study drug or the subject's EOS visit, whichever is later.
Description: In the first treated eye all events/conditions will be captured as an AE as treatment continues from the preceding study.
Arm/Group | Drug QR-110
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug QR-110 (N=9)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug QR-110 (N=9)
Cataract (Eye disorders) | 1
Cataract cortical (Eye disorders) | 1
Cataract subcapsular (Eye disorders) | 2
Conjunctival haemorrhage (Eye disorders) | 2
Cystoid macular oedema (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Lenticular opacities (Eye disorders) | 2
Posterior capsule opacification (Eye disorders) | 3
Retinal cyst (Eye disorders) | 1
Retinal degeneration (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 3
Infections and infestations (Eye disorders) | 1
Blebitis (Infections and infestations) | 1
Posterior lens capsulotomy (Surgical and medical procedures) | 1
Fatigue (General disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Cystitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Coronavirus test positive (Investigations) | 1
Headache (Nervous system disorders) | 1
Petit mal epilepsy (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Dermabrasion (Surgical and medical procedures) | 1
Wisdom teeth removal (Surgical and medical procedures) | 1
Diplopia (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution shall be free to publish, present, or use any Data and results arising out of its performance of the protocol. At least 30 days prior to submission for publication, institution shall submit to Sponsor for review and comment any proposed oral or written publication. Institution will consider any such comments in good faith but is under no obligation to incorporate Sponsor's suggestions. The review period for abstracts or poster presentations shall be 30 days.

DOCUMENTS (2):
  • Study Protocol (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT03913130/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT03913130/SAP_001.pdf